CLINICAL TRIAL: NCT04410354
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Oral Merimepodib in Combination With Intravenous Remdesivir in Adult Patients With Advanced Coronavirus Disease 2019 (COVID-19)
Brief Title: Study of Merimepodib in Combination With Remdesivir in Adult Patients With Advanced COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failure to meet primary endpoint
Sponsor: ViralClear Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VC-02-01
Record Dates: First submitted 2020-04-28; First posted 2020-06-01 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: COVID-19
Keywords: Coronavirus; Advanced Coronavirus Disease 2019; SARS-Cov-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — N-3-(3-(3-methoxy-4-oxazol-5-ylphenyl)ureido)benzylcarbamic acid tetrahydrofuran-3-yl ester; remdesivir

STUDY DESIGN:
Intervention Model Description: Eligible study subjects will be randomized 1:1 to receive oral administration of study drug or placebo. Both treatment arms will also receive remdesivir.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Pharmacy prepares medications that are coded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MMPD + remdesivir (Active Comparator): Study subjects will receive MMPD oral solution 3 times per day for 10 days unless discontinued early. Study subjects will also receive remdesivir infusion once a day for 5 days. If a subject does not demonstrate clinical improvement, remdesivir treatment may be extended for up to 5 additional days (for a total of up to 10 days).
  Interventions: Drug: Merimepodib; Drug: Remdesivir
- Placebo + remdesivir (Placebo Comparator): Study subjects will receive matching placebo oral solution 3 times per day for 10 days unless discontinued early. Study subjects will also receive remdesivir infusion once a day for 5 days. If a subject does not demonstrate clinical improvement, remdesivir treatment may be extended for up to 5 additional days (for a total of up to 10 days).
  Interventions: Drug: Matching Placebo; Drug: Remdesivir

INTERVENTIONS:
Drug: Merimepodib — 400 mg (total daily dose of 1200 mg) for 10 days
  Other Names: VX-497
  Arms: MMPD + remdesivir
Drug: Matching Placebo — 0 mg (total daily dose of 0 mg) for 10 days
  Arms: Placebo + remdesivir
Drug: Remdesivir — 200 mg loading dose on Day 0 followed by 100 mg daily dose for 4 days. If a subject does not demonstrate clinical improvement, 100 mg daily dose may be extended for up to 5 additional days (for a total of up to 10 days)

SUMMARY:
The purpose of this study is to assess the safety and efficacy of merimepodib (MMPD) oral solution when administered in combination with remdesivir in adult patients with advanced COVID-19.

DETAILED DESCRIPTION:
This phase 2 randomized, double-blind, placebo-controlled study will enroll approximately 80 adult patients with advanced coronavirus disease 2019 (COVID-19). Approximately 80 patients will be randomized 1:1 to receive oral administration of MMPD + remdesivir or placebo + remdesivir. The first 40 patients will have a score of 3 or 4 on the National Institute of Allergy and Infectious Disease (NIAID) 8-point ordinal scale and at least one of the following: fever, cough, sore throat, malaise, headache, muscle pain, shortness of breath at rest or with exertion, confusion or symptoms of severe lower respiratory symptoms; the final 40 patients will have a score of 3 on the NIAID scale.

Study subjects will undergo screening evaluations prior to the first dose of study drug. Study drug treatment (MMPD or placebo) will continue for 10 days, unless the patient is discharged from the hospital before completing the 10-day randomized treatment period. Both treatment arms will also receive remdesivir per the Emergency Use Authorization labeling. Evaluations will be performed on Days 0-10 and every day thereafter until the subject no longer requires any form of respiratory support or they reach the last planned day of in-person study assessments and still require respiratory support. The final in-person study evaluations will be performed 4 weeks after completion of study drug (MMPD or placebo) treatment (Day 37). The final study evaluation will be a telephone call on Day 56.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Confirmed SARS-CoV-2 viral infection
* Advanced COVID-19 with score of 3 or 4 on NIAID scale (first 40 patients) or score of 3 on NIAID scale (last 40 patient
* Has at least one of the following: fever, cough, sore throat, malaise, headache, muscle pain, shortness of breath, confusion or severe lower respiratory symptoms
* Off antiviral medications at least 24 hours prior to first dose of study drug (except for remdesivir)
* Able to provide consent
* Agree to appropriate methods of contraception

Exclusion Criteria:

* In critical condition or has ARDS
* On invasive mechanical ventilation or ECMO
* Bacterial or fungal infection
* Pregnant or lactating (women)
* ALT >5x ULN, bilirubin >2x ULN, INR outside of normal limits at screening
* eGFR <30 mL/min
* Clinically relevant serious co-morbid medical conditions
* Treatment with any immunosuppressive therapy within 30 days prior to screening
* Treatment with another investigational drug within 30 days or 5 half-lives of drug prior to screening
* Prior treatment with the study drug (MMPD) or treatment with remdesivir more than 24 hours prior to the first randomized dose of study drug
* Known hypersensitivity to the inactive ingredients in the study drug (MMPD or placebo) or any ingredient of remdesivir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects not hospitalized or, if hospitalized, free of respiratory failure | Day 0 to Day 28
  Proportion of subjects alive at Day 28 who are not hospitalized or if hospitalized are free of respiratory failure
Adverse Events | Day 0 to Day 56
  Number of Adverse Events (AEs) and number & percentage of subjects experiencing AEs after administration of the first dose of study drug

SECONDARY OUTCOMES:
National Institute of Allergy and Infectious Disease (NIAID) 8-Point Ordinal Scale | Day 0 to Day 28
  Change in NIAID 8-point ordinal scale, where 1=Death and 8=Not hospitalized, no limitations on activities
Temperature | Day 0 to Day 37
  Duration of fever
Death | Day 0 to Day 56
  Number of deaths
Mechanical ventilation | Day 0 to Day 56
  Need and duration of mechanical ventilation
Vasopressor Support | Day 0 to Day 56
  Duration of vasopressor support
Oxygen Therapy | Day 0 to Day 37
  Duration of oxygen therapy via mechanical ventilation, face mask or nasal cannula
Cessation of Viral Shedding | Day 0 to Day 37
  Time to cessation of viral shedding based on absence of SARS-CoV-2 in a PCR based COVID-19 test
Change in Oxygen Saturation/Fraction of Inspired Oxygen | Day 0 to Day 37
  Change in SpO2/FiO2

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Badley, MD, Study Director — Mayo Clinic
Locations (10):
- United States (10):
  - Mayo Clinic in Arizona, Phoenix, Arizona
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Atlantic Health System / Morristown Medical Center, Morristown, New Jersey
  - Atlantic Health System / Overlook Medical Center, Summit, New Jersey
  - St. David's South Austin Medical Center, Austin, Texas
  - St. David's Medical Center, Austin, Texas
  - HCA Houston Healthcare Medical Center, Houston, Texas
  - HCA Houston Healthcare Mainland, Texas City, Texas

IPD SHARING:
Plan to Share IPD: No